CLINICAL TRIAL: NCT07280676
Title: The Effect of Cosmetic Formulations on the Appearance of Gray Hair
Brief Title: The Effect of Cosmetic Formulations on the Appearance of Grey Hair.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Comprehensive Research Group, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMN-BIO-4402
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Hair Graying
Keywords: Hair appearance; Hair graying
MeSH Terms: interventions — RNA, U82 small nucleolar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cosmetic product U82 (Experimental): Cosmetic scalp leave on product to be used once daily on the whole scalp for 6 months.
  Interventions: Other: U82
- Cosmetic product Z63 (Experimental): Cosmetic scalp leave on product to be used once daily on the whole scalp for 6 months.
  Interventions: Other: Z63

INTERVENTIONS:
Other: U82 — Cosmetic scalp leave on product
  Arms: Cosmetic product U82
Other: Z63 — Cosmetic scalp leave on product
  Arms: Cosmetic product Z63

SUMMARY:
This study is a 6-month (180 days) single-center, double blind study designed to explore the effect of two cosmetic products on the appearance of gray hair.

DETAILED DESCRIPTION:
This is a randomised, double blind, whole head study designed to evaluate the effect of two cosmetic leave on treatments on the appearance of gray hair. This study will accept up to 190 participants per cell (380 participants overall) who meet the inclusion/exclusion criteria to ensure that at least 150 participants per cell complete the study. Participants will be randomised to receive one of the two cosmetic hair products. The products will be applied to the whole scalp using a defined protocol.

If accepted onto the study, participants will be provided with marketed shampoo and conditioner products for use throughout the study.

Visual and instrumental assessments of hair color will be conducted throughout the duration of the study (6 months/180 days). Non-invasive skin surface samples will be collected at baseline, day 90 and day 180 for evaluation of target proteins and untargeted proteomic analysis of scalp and hair health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Female or Male between the ages of 25 and 60 years old, both inclusive at the time of consent.
* Of any race and ethnicity.
* Able to read and understand all study instructions and any other relevant study documents and understand the test procedures (in English) and able to provide a free decision about participating in the study.
* Has 15 - 35% naturally gray hair
* Available to come to all study visits.

Exclusion Criteria:

* Individuals with any relevant past or present medical history which may affect the study results or may lead to increased risk to the participant in the judgement of the Investigator or designee, including a history of cancer, insulin-dependent diabetes, acute or chronic renal insufficiency, chronic inflammatory disorders (arthritis, osteoarthritis, inflammatory bowel disease, colitis, etc.), asthma (not including exercise-induced asthma), epilepsy, uncontrolled hyperthyroidism, or uncontrolled hypothyroidism. Participants who have well controlled hyperthyroidism and hypothyroidism (stable medication for greater than 6 months) will be permitted.
* Pattern hair loss (Savin ≥ 2 for females, or Hamilton-Norwood ≥IV & excluding vertex hair loss for males) or any history of hair loss for medical reasons, including, but not limited to, alopecia areata, alopecia universalis, alopecia totalis or telogen effluvium.
* Individuals that are sensitive/allergic to any of the ingredients in any of the test products adhesives, tattoo pigments/ink, or metals used in needles (i.e., chromium or nickel).
* Individuals with an immunological disorder or bloodborne disease (e.g. HIV, HBC, AIDS, multiple sclerosis, Crohn's disease, rheumatoid arthritis) or currently using oral or systemic immunosuppressive medications and biologics (e.g., azathioprine, belimumab, Cimzia®, Cosentyx®, cyclophosphamide, cyclosporine, Enbrel®, Humira®, Imuran®, Kineret®, mycophenolate mofetil, methotrexate, Orencia®, prednisone, Remicade®, Rituxan®, Siliq™, Simponi®, Stelara®, Taltz®) and/or undergoing radiation or chemotherapy as determined by study documentation.
* Individuals having started a long-term medication within the last 6 months or have changed brand, manufacture, or dosage of a long-term medication.
* Individuals currently using or having regularly used corticosteroids (known as steroids), systemically or topically, topically anywhere on the body, except nasal, and/or ocular use is acceptable within the past 4 weeks (including but not limited to betamethasone, clobetasol, desoximetasone, diflorasone, fluocinonide, fluticasone, mometasone, halcinonide, and halobetasol) (see list in Appendix 8)
* Individuals currently taking any other medications which, in the opinion of the Investigator or designee, may interfere with the study (e.g. prescription anti-inflammatory drugs, anticoagulants, etc.).
* Individuals with hemophilia, anemia, or any other blood clotting disorder.
* Individuals who have a history of systemic granulomatous diseases, active or inactive, (e.g., sarcoidosis, Wegener's granulomatosis, tuberculosis) or connective tissue diseases (e.g., lupus, dermatomyositis).
* Individuals who are involved in any aspect of administration or an employee of Sponsor or testing facility.
* Individuals currently used/taking or have used/taken within the last 3 months any topical or ingestible anti-gray hair or hair growth supplements/treatments (examples: Arey: Not Today, Anti-gray hair supplements, Heyhair: Gray Escape Advanced Anti-Gray Hair Growth Supplements, Vegamour: GRO Ageless Gray Delay Hair Supplements, Elon Essentials, R3 Extra Strength etc.).

The Investigator may exclude participants for other conditions, factors, or medications that they believe may affect the response of the skin or the interpretation of the test results.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Visual assessment of percent gray hair | 0 - 6 months
  Percent gray hair assessed over the whole head by expert assessor
Image analysis of appearance of gray hair | 0 - 6 months
  Image analysis of global photographs of the head

SECONDARY OUTCOMES:
Image analysis of individual hair fibre color | 0 - 6 months
  Image analysis of macro photographs of selected areas of the scalp
Consumer perception of scalp and hair condition and hair grayness | 0 - 6 months
  Questionnaires

OTHER OUTCOMES:
Proteomic analysis of scalp surface proteins associated with scalp and hair health | 0 - 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Research Group, Inc., Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No